CLINICAL TRIAL: NCT06562764
Title: Role of Pharmaceutical Pictograms in Disease Management: A Mix Method Study of Various Stakeholders in Pakistan
Brief Title: To Evaluate Newly Developed Pictogram Cards and Their Utility in Improving Inhaler Techniques in Asthmatic Patients
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Islamia University of Bahawalpur (Other)
Responsible Party: Principal Investigator, Kanza Arshad, PhD Scholar, Islamia University of Bahawalpur
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 668/AS&R
Record Dates: First submitted 2024-07-27; First posted 2024-08-20 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-08

CONDITIONS: Asthma
Keywords: Pictograms; MDI; DPI; Inhaler; Pictogram cards; Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Intervention Model Description: A parallel study is a type of clinical study in which two or more groups of participants receive different interventions. Participants are assigned to one of the treatment arms at the beginning of the trial and continue in that arm throughout the length of the trial.
Masking Description: An open-label trial, or open trial, is a type of clinical trial in which information is not withheld from trial participants.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Controlled (No Intervention): The control group is the set of subjects that do not receive the intervention in a study.
- Counselling by the Trained Pharmacist (Experimental): The intervention group 1 is the set of subjects that receive the "counseling intervention" in a study.
  Interventions: Other: Counselling by the Trained Pharmacist
- Counselling and Pictograms (Experimental): Intervention group 2 consists of the subjects who receive the "counseling and pictogram intervention" in a study.
  Interventions: Other: Pictograms Cards and Counselling by the Trained Pharmacist

INTERVENTIONS:
Other: Counselling by the Trained Pharmacist — The intervention group 1 is verbally counselled about the proper use of their inhaler devices.
  Arms: Counselling by the Trained Pharmacist
Other: Pictograms Cards and Counselling by the Trained Pharmacist — The investigator developed pictogram cards for the use of inhalers (MDI and DPI) and pictogram cards are attached to the inhalers of patients in the intervention group with counselling by the trained pharmacist.
  Arms: Counselling and Pictograms

SUMMARY:
To evaluate newly developed pictogram cards and their utility in improving inhaler techniques in asthmatic patients.

DETAILED DESCRIPTION:
A prospective, open-label, randomized controlled clinical study. For this purpose, pictogram cards are designed for Metered Dose Inhalers (MDI) and Dry Powder Inhalers (DPI).

The pictogram labels are designed and printed in colors with Urdu language and then attached to the inhaler devices as cards. The demographic, clinical, and medical data are collected from the patients and their medical files. Moreover, the different clinical measures are also evaluated in the recruited patients.

ELIGIBILITY:
Inclusion Criteria:

* Asthmatic Patients, should take inhalers regularly for at least 3 months and come personally for re-fill.

Exclusion Criteria:

* Coexistence of other chronic respiratory conditions.
* Those who were difficult to communicate.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 320 (Actual)
Dates: Start 2024-05-10 (Actual); Primary Completion 2024-06-20 (Actual); Study Completion 2024-08-25 (Estimated)

PRIMARY OUTCOMES:
Proper/Improper use of inhaler | 12 weeks
  Determine the proper/improper use of inhaler via checklist. The dichotomous primary endpoint (Proper inhaler technique/ Improper Inhaler Technique). A participant is categorized as having proper inhaler technique if the score was 7/7 and improper technique if the score was < 7.

SECONDARY OUTCOMES:
Determine the adherence via a validated tool named the Medication Adherence Report Scale (MARS-5). | 12 weeks
  Adherence is the extent to which a person's behavior- taking medication, following a diet, and/or executing lifestyle changes- corresponds with the agreed recommendations from a healthcare provider. The adherence is measured via a validated tool named the Medication Adherence Report Scale (MARS-5). MARS-5 shows promise as a self-report tool for measuring patients' reports of their medication use across various illnesses. The score ranges from 5 to 25, where a higher MARS-5 score indicates higher self-reported adherence.
Determine the Asthma Control in the asthmatic patients via ACT questionnaire. | 12 weeks
  Asthma control is determined via ACT questionnaire. ACT scores range from 5-25 for the adult test and 0-27 for the child test. The higher the score, the better the asthma control. In both tests, a score of 20 or higher suggests your asthma is probably under control.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Muhammad Atif, PhD, Study Director — The Islamia University of Bahawalpur
Locations (1):
- The Islamia University of Bahawalpur, Chak Four Hundred Fifty-four, Bahawalpur, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
The IPD collected during the trial allowed by the research investigator, after deidentification.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: Immediately after publication and no end date.
Access Criteria: Researchers who provide the methodologically sound proposal.